CLINICAL TRIAL: NCT00144664
Title: An Open-Label, Phase III Study to Evaluate the Efficacy, Safety and PK of MRA in Patients With pJIA
Brief Title: Study of MRA for Polyarticular Juvenile Idiopathic Arthritis (pJIA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRA318JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Systemic Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): MRA(Tocilizumab)
  Interventions: Drug: MRA(Tocilizumab)

INTERVENTIONS:
Drug: MRA(Tocilizumab)

SUMMARY:
This is an open-label, Phase III study to evaluate the efficacy, safety and PK of MRA in patients with pJIA.

ELIGIBILITY:
Inclusion criteria

* Patients who are diagnosed with rheumatoid factor (RF) positive or negative polyarthritic or oligoarthritic JIA according to the ILAR standards (1997)
* Patients aged at least 2 years old and less than 20.
* Patients aged less than 16 years old at time of onset

Exclusion criteria

* Patients with Class IV Steinbrocker functional disorder at evaluation within 2 weeks before initiation of treatment with the investigational product
* Patients who have been treated for the underlying disease with a biological agent, such as infliximab or etanercept, within 12 weeks before initiation of treatment with the investigational product

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2004-11; Primary Completion 2005-04 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Efficacy:Percentage of patients showing 30% improvement in the JIA core set on LOBS | whole period
Safety:Incidence and severity of adverse events and adverse drug reactions | whole period
Pharmacokinetics:The Cmax, trough values, AUC, Kel, CL, Vd, Vdss, and t1/2 for serum MRA concentration | whole period

SECONDARY OUTCOMES:
Efficacy:The time course of the percentage of patients showing 30%, 50%, and 70% improvement in the JIA core set, each evaluation endpoint in the JIA core set, CRP, pain up to LOBS | whole period

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Kakehi, Study Director — Chugai Pharmaceutical